CLINICAL TRIAL: NCT02421380
Title: Characterization of Hyperpolarized Pyruvate MRI Reproducibility
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 14-205
Record Dates: First submitted 2015-04-13; First posted 2015-04-20 (Estimated); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Malignant Solid Tumors
Keywords: Hyperpolarized Pyruvate; MRI; 14-205

ARMS (1):
- Hyperpolarized Pyruvate MRI Reproducibility (Experimental): This is a reproducibility study of hyperpolarized [1-13C] pyruvate MRI in patients with solid tumors. A total of 100 patients will be enrolled, 50 of whom will be imaged using 1D MR spectroscopy and the other 50 with 3D imaging sequence.
  Interventions: Drug: Hyperpolarized Pyruvate

INTERVENTIONS:
Drug: Hyperpolarized Pyruvate

SUMMARY:
The purpose of the study is to test a new approach to see if the test results can be reproduced each time the Magnetic resonance imaging (MRI) is done for an individual patient. The study will explore the use of an imaging agent called hyperpolarized [1-13C] pyruvate (HP) with MRI scans. (MRI) is a technique that takes pictures of the body's organs using a magnetic field and radiofrequency waves that cannot be felt. In order to accomplish the goal of the study the patient will have two hyperpolarized MRI scans to assess if scans can be reproduced. The hyperpolarized MRI scans will be compared with the pathological results of the surgery to see if the hyperpolarized MRI provides additional information regarding disease metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Patients with history of histologically-confirmed malignant solid tumor (histology confirmed by MSKCC Department of Pathology.) NOTE: An exception will be made for patients with brain lesions. Patients identified by a radiologist to have a brain lesion with high suspicion for neoplasm given MRI features will be enrolled, prior to histological confirmation.
* Disease measurable or evaluable as defined by RECIST 1.1, a mass of greater than 1cm in the long axis and/or other tumor response criteria from an MSKCC IRB-approved clinical research protocol. NOTE: Study patients do not need to be participating in an MSKCC approved clinical trial prior to study recruitment.
* Negative serum or urine pregnancy test for female patients of childbearing age and potential (as defined by MSKCC Standards & Guidelines), from assays obtained < 2 weeks prior to study enrollment.
* This study will include only patients with sarcoma, prostate, breast, brain, metastatic or pancreatic cancer. In the future other patient groups may be included through amendment of this protocol.

Exclusion Criteria:

* Inability or refusal to have at least one peripheral intravenous line for intravenous access (as applicable to the day of [1-13C] pyruvate injection)
* Breast-feeding
* Refusal or inability to tolerate the scanning procedure (e.g., due to claustrophobia)
* Hepatic: from assays obtained within 3-4 weeks prior to study enrollment. For each patient, the upper limit of normal (ULN) value for a particular assay will be defined by the normal reference values of the laboratory that performed the assay
* Bilirubin > 1.5 x (ULN)
* AST/ALT >2.5 x ULN
* Albumin < 3 g/dl
* GGT > 2.5 x ULN if Alkaline phosphatase > 2.5 x ULN.
* Renal: Creatinine >1.5 x ULN or creatinine clearance < 60 mL/min, from assays obtained within 3-4 weeks prior to study enrollment
* Acute major illness (e.g., unstable cardiovascular condition, etc.)
* Standard MRI exclusion criteria will also be applied, including pacemakers and metal clips located in the patient.

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Estimated)
Dates: Start 2015-04 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
validate HP MRI at MSKCC (are the scans able to be reproduced) | 1 year
  The imaging will include standard T2-weighted, diffusion-weighted (DW), dynamic contrast-enhanced (DCE) and 1H MR spectroscopic imaging, depending on the solid tumor type. This multi-parametric data will be used to delineate the tumor as well as compare to HP MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Kayvan Keshari, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - Memorial Sloan Kettering Bergen (Consent only ), Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York

REFERENCES:
- [Derived] Granlund KL, Tee SS, Vargas HA, Lyashchenko SK, Reznik E, Fine S, Laudone V, Eastham JA, Touijer KA, Reuter VE, Gonen M, Sosa RE, Nicholson D, Guo YW, Chen AP, Tropp J, Robb F, Hricak H, Keshari KR. Hyperpolarized MRI of Human Prostate Cancer Reveals Increased Lactate with Tumor Grade Driven by Monocarboxylate Transporter 1. Cell Metab. 2020 Jan 7;31(1):105-114.e3. doi: 10.1016/j.cmet.2019.08.024. Epub 2019 Sep 26. PMID 31564440
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/